CLINICAL TRIAL: NCT03635983
Title: A Phase 3, Randomized, Open-label Study of NKTR-214 Combined With Nivolumab Versus Nivolumab in Participants With Previously Untreated Unresectable or Metastatic Melanoma
Brief Title: A Study of NKTR-214 Combined With Nivolumab vs Nivolumab Alone in Participants With Previously Untreated Inoperable or Metastatic Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA045-001; 2018-001423-40 (EudraCT Number); 17-214-08 (Other: Nektar Therapeutics)
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Melanoma
Keywords: NKTR-214; Nivolumab; Immunotherapy; bempegaldesleukin (BEMPEG: NKTR-214)
MeSH Terms: conditions — Melanoma | interventions — bempegaldesleukin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination (Experimental): NKTR-214 + Nivolumab
  Interventions: Biological: NKTR-214; Biological: Nivolumab
- Monotherapy (Experimental): Nivolumab
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: NKTR-214 — Specified dose on specified days
  Other Names: Bempegaldesleukin; BMS-986321
  Arms: Combination
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558

SUMMARY:
The purpose of the study is to test the effectiveness (how well the drug works), safety, and tolerability of the investigational drug called NKTR-214, when combined with nivolumab versus nivolumab given alone in participants with previously untreated melanoma skin cancer that is either unable to be surgically removed or has spread

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1 (adults 18 years or older)/Lansky Performance Score ≥ 80% (minors ages 12-17 only)
* Histologically confirmed stage III (unresectable) or stage IV melanoma
* Treatment-naive participants (ie, no prior systemic anticancer therapy for unresectable or metastatic melanoma) with the exception of prior adjuvant and/or neoadjuvant treatment for melanoma with approved agents

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases
* Uveal melanoma
* Participants with an active, known or suspected autoimmune disease

Other protocol defined inclusion/exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 783 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2024-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (167):
- United States (24):
  - Local Institution - 0187, Tucson, Arizona
  - Local Institution - 0014, La Jolla, California
  - Local Institution - 0122, Stanford, California
  - Local Institution - 0051, Aurora, Colorado
  - Local Institution - 0065, New Haven, Connecticut
  - Local Institution - 0153, Miami, Florida
  - Local Institution - 0017, Miami Beach, Florida
  - Local Institution - 0112, Tampa, Florida
  - Local Institution - 0012, Atlanta, Georgia
  - Local Institution - 0019, Louisville, Kentucky
  - Local Institution - 0018, Boston, Massachusetts
  - Local Institution - 0188, Ann Arbor, Michigan
  - Local Institution - 0186, Fridley, Minnesota
  - Local Institution - 0135, St Louis, Missouri
  - Local Institution - 0016, Hackensack, New Jersey
  - Local Institution - 0185, New Brunswick, New Jersey
  - Local Institution - 0141, New York, New York
  - Local Institution - 0037, Cleveland, Ohio
  - Local Institution - 0011, Portland, Oregon
  - Local Institution - 0013, Portland, Oregon
  - St. Luke's Hospital & Health Network, Easton, Pennsylvania
  - Local Institution - 0015, Philadelphia, Pennsylvania
  - Local Institution - 0001, Houston, Texas
  - Local Institution - 0064, Fairfax, Virginia
- Argentina (5):
  - Local Institution - 0109, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0107, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0183, Buenos Aires, Distrito Federal
  - Local Institution - 0108, CABA
  - Local Institution - 0157, Córdoba
- Australia (10):
  - Local Institution - 0146, Coffs Harbour, New South Wales
  - Local Institution - 0053, North Sydney, New South Wales
  - Local Institution - 0058, Cairns, Queensland
  - Local Institution, Greenslopes, Queensland
  - Local Institution - 0056, Woolloongabba, Queensland
  - Local Institution - 0172, Elizabeth Vale, South Australia
  - Local Institution - 0054, Melbourne, Victoria
  - Local Institution - 0143, Melbourne, Victoria
  - Local Institution - 0057, Nedlands, Western Australia
  - Local Institution - 0097, Nedlands, Western Australia
- Austria (3):
  - Local Institution - 0034, Graz
  - Local Institution - 0035, Salzburg
  - Local Institution - 0033, Vienna
- Belgium (3):
  - Local Institution - 0083, Brussels
  - Local Institution - 0084, Hasselt
  - Local Institution - 0085, Leuven
- Brazil (8):
  - Local Institution - 0168, Fortaleza, Ceará
  - Local Institution - 0125, Belo Horizonte, Minas Gerais
  - Local Institution - 0124, Ijuí, Rio Grande do Sul
  - Local Institution - 0127, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0171, Itajaí, Santa Catarina
  - Local Institution - 0126, Barretos, São Paulo
  - Local Institution - 0182, Rio de Janeiro
  - Local Institution - 0169, São Paulo
- Canada (7):
  - Local Institution - 0068, Abbotsford, British Columbia
  - Local Institution - 0139, St. John's, Newfoundland and Labrador
  - Local Institution - 0066, Hamilton, Ontario
  - Local Institution - 0067, Kitchener, Ontario
  - Local Institution - 0041, Toronto, Ontario
  - Local Institution, Québec, Quebec
  - Local Institution - 0121, Edmonton
- Chile (2):
  - Local Institution - 0174, Recoleta, Santiago Metropolitan
  - Local Institution - 0173, Santiago, Santiago Metropolitan
- Czechia (4):
  - Local Institution - 0094, Brno
  - Local Institution - 0093, Hradec Králové
  - Local Institution - 0091, Prague
  - Local Institution - 0092, Prague
- Finland (3):
  - Local Institution - 0166, Tampere, Oulun Lääni
  - Local Institution - 0167, KYS
  - Local Institution - 0165, Turku
- France (11):
  - Centre Hospitalier Universitaire de Bordeaux Hospital Saint Andre, Bordeaux
  - Hopital Claude Huriez, Lille
  - Hopital Saint Eloi, Montpellier
  - Local Institution - 0003, Nantes
  - Local Institution - 0155, Nice
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Charles Nicolle, Rouen
  - Local Institution - 0009, Saint-Priest-en-Jarez
  - Local Institution - 0002, Toulouse
  - Institute Gustave Roussy, Villejuif
- Germany (15):
  - Local Institution - 0031, Buxtehude
  - Local Institution - 0029, Dresden
  - Local Institution - 0192, Erfurt
  - Local Institution - 0026, Essen
  - Local Institution - 0030, Göttingen
  - Local Institution - 0023, Hamburg
  - Local Institution - 0024, Hanover
  - Local Institution - 0020, Heidelberg
  - Local Institution - 0028, Kiel
  - Local Institution - 0022, Leipzig
  - Local Institution - 0021, München
  - Local Institution - 0027, Münster
  - Local Institution - 0060, Regensburg
  - Local Institution - 0025, Tübingen
  - Local Institution - 0032, Würzburg
- Greece (3):
  - Local Institution - 0038, Athens
  - Local Institution - 0039, Neo Faliro
  - Local Institution - 0040, Thessaloniki
- Ireland (4):
  - Local Institution - 0136, Wilton, CORK
  - Local Institution - 0129, Dublin, Dublin
  - Local Institution - 0128, Dublin
  - Local Institution - 0130, Dublin
- Israel (3):
  - Local Institution - 0098, Beersheba
  - Local Institution - 0088, Jerusalem
  - Local Institution - 0089, Ramat Gan
- Italy (10):
  - Local Institution - 0045, Milan, Lombardy
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Local Institution - 0044, Bari
  - ASST Papa Giovanni XXIII, Bergamo
  - Local Institution - 0113, Meldola (FC)
  - IRCCS Istituto Nazionale Tumori Milano, Milan
  - Local Institution - 0043, Napoli
  - Istituto Oncologico Veneto IOV, Padua
  - Local Institution - 0042, Siena
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Torino
- Mexico (7):
  - Local Institution - 0176, Zapopan, Jalisco
  - Local Institution - 0175, Mexico City, Mexico City
  - Local Institution - 0177, Monterrey, Nuevo León
  - Local Institution - 0180, Monterrey, Nuevo León
  - Local Institution - 0178, Cancún, Quintana Roo
  - Local Institution - 0179, Puebla City
  - Local Institution - 0181, San Luis Potosí City
- Netherlands (5):
  - Local Institution - 0101, Amsterdam
  - Local Institution - 0102, Amsterdam
  - Local Institution - 0099, Leiden
  - Local Institution - 0100, Nijmegen
  - Local Institution - 0147, Untrecht
- New Zealand (3):
  - Local Institution - 0159, Auckland
  - Local Institution - 0063, Christchurch
  - Local Institution - 0062, Wellington
- Poland (2):
  - Local Institution - 0152, Bydgoszcz
  - Local Institution - 0090, Warsaw
- Portugal (2):
  - Local Institution - 0134, Lisbon
  - Local Institution - 0133, Porto
- Romania (4):
  - Local Institution - 0162, Bucharest
  - Local Institution - 0070, Cluj-Napoca
  - Local Institution - 0071, Craiova
  - Local Institution - 0120, Floreşti
- Russia (4):
  - Local Institution - 0149, Krasnoyarsk
  - Local Institution - 0086, Moscow
  - Local Institution - 0111, Moscow
  - Local Institution - 0148, Moscow
- Spain (9):
  - Local Institution - 0116, Barcelona
  - Local Institution - 0115, Barcelona
  - Local Institution - 0123, Córdoba
  - Local Institution - 0190, Doniostia - San Sebastian
  - Local Institution, Donostia / San Sebastian
  - Local Institution - 0118, Jaén
  - Local Institution - 0114, Madrid
  - Local Institution - 0119, Santiago Compostela
  - Local Institution - 0117, Valencia
- Sweden (2):
  - Local Institution - 0163, Gothenburg
  - Local Institution - 0164, Lund
- Switzerland (3):
  - Local Institution - 0104, Bern
  - Local Institution - 0105, Lausanne
  - Local Institution - 0036, Zurich
- United Kingdom (11):
  - Local Institution - 0132, Southampton, Hampshire
  - Local Institution, Edinburgh, Midlothian
  - Local Institution - 0131, Sutton, Surrey
  - Local Institution - 0078, Belfast
  - Local Institution - 0076, Cambridge
  - Local Institution - 0079, Cottingham
  - Local Institution - 0137, Liverpool
  - Local Institution - 0077, London
  - Local Institution - 0074, London
  - Local Institution - 0075, Manchester
  - Local Institution - 0142, Tauton

REFERENCES:
- [Derived] Diab A, Gogas H, Sandhu S, Long GV, Ascierto PA, Larkin J, Sznol M, Franke F, Ciuleanu TE, Pereira C, Munoz Couselo E, Bronzon Damian F, Schenker M, Perfetti A, Lebbe C, Quereux G, Meier F, Curti BD, Rojas C, Arriaga Y, Yang H, Zhou M, Ravimohan S, Statkevich P, Tagliaferri MA, Khushalani NI. Bempegaldesleukin Plus Nivolumab in Untreated Advanced Melanoma: The Open-Label, Phase III PIVOT IO 001 Trial Results. J Clin Oncol. 2023 Oct 20;41(30):4756-4767. doi: 10.1200/JCO.23.00172. Epub 2023 Aug 31. PMID 37651676
- [Derived] Khushalani NI, Diab A, Ascierto PA, Larkin J, Sandhu S, Sznol M, Koon HB, Jarkowski A, Zhou M, Statkevich P, Geese WJ, Long GV. Bempegaldesleukin plus nivolumab in untreated, unresectable or metastatic melanoma: Phase III PIVOT IO 001 study design. Future Oncol. 2020 Oct;16(28):2165-2175. doi: 10.2217/fon-2020-0351. Epub 2020 Jul 29. PMID 32723187
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Bempegaldesleukin + Nivolumab: Bempegaldesleukin 0.006 mg/kg IV every 3 weeks + Nivolumab 360 mg IV every 3 weeks
- Nivolumab: Nivolumab 360 mg IV every 3 weeks
Period: Pre-Treatment Period
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Started (Started=randomized) | 391 | 392
Completed (Completed=treated) | 388 | 382
Not Completed | 3 | 10
Not completed — Withdrawal by Subject | 0 | 7
Not completed — Participant no longer meets study criteria | 1 | 0
Not completed — Other reasons | 0 | 1
Not completed — Disease Progression | 0 | 1
Not completed — Adverse Event unrelated to Study drug | 2 | 1
Period: Treatment Period
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Started (Started=treated) | 388 | 382
Completed | 82 | 96
Not Completed | 306 | 286
Not completed — Participant request to discontinue Study treatment | 6 | 7
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Death | 3 | 5
Not completed — Poor/Non-compliance | 2 | 1
Not completed — Participant no longer meets Study criteria | 1 | 4
Not completed — Other reasons | 7 | 4
Not completed — Disease progression | 230 | 201
Not completed — Study drug toxicity | 35 | 36
Not completed — Adverse event unrelated to Study drug | 15 | 15
Not completed — Maximum clinical benefit | 3 | 5
Not completed — Administrative reason by the sponsor | 1 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab | Total
Number analyzed (Participants) | 391 | 392 | 783
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (13.2) | 60.4 (13.5) | 60.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 163 | 325
  Male | 229 | 229 | 458
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 81 | 73 | 154
  Not Hispanic or Latino | 165 | 153 | 318
  Unknown or Not Reported | 145 | 166 | 311
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 379 | 379 | 758
  Black or African American | 2 | 4 | 6
  Asian | 1 | 0 | 1
  American Indian or Alaska Native | 5 | 2 | 7
  Other | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Blinded Independent Central Review (BICR)
Description: ORR is defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR) using RECIST v 1.1 per blinded independent central review (BICR) assessment. CR=Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From date of randomization to disease progression (Up to 37 months)
Population: All randomized participants with at least 6 months of follow-up at the time point of the final ORR analysis. A follow-up time is defined as the time between randomization date and clinical data cut-off date.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 271 | 272
Percentage of participants | 27.7 [22.4 to 33.4] | 36.0 [30.3 to 42.0]
Statistical Analysis 1: Comparison: Bempegaldesleukin + Nivolumab vs Nivolumab; Bempegaldesleukin+Nivolumab over Nivolumab; Test type: Superiority; p = 0.0311, Stratified Cochran-Mantel-Haenszel; two-sided; Estimate of Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.45 to 0.96] — Strata adjusted odds ratio (NKTR-214 + Nivolumab over Nivolumab) using Mantel-Haenszel method

2. Primary Outcome: Progression-free Survival (PFS) Per Blinded Independent Central Review (BICR)
Description: PFS is defined as the time between the date of randomization and the first date of documented tumor progression using RECIST v 1.1 per blinded independent central review (BICR), or death due to any cause, whichever comes first. Progressive disease (PD)=At least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From date of randomization to disease progression, or death, whichever comes first (Up to 37 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 391 | 392
Months | 4.17 [3.52 to 5.55] | 4.99 [4.14 to 7.82]
Statistical Analysis 1: Comparison: Bempegaldesleukin + Nivolumab vs Nivolumab; Test type: Superiority; p = 0.3988, Log Rank — Log-rank stratified 2-sided. Boundary for statistical significance p-value < 0.03; Hazard Ratio (HR) = 1.09, 95% CI [0.89 to 1.33] — Stratified Cox proportional hazard model. Hazard Ratio is NKTR-214 + Nivolumab over Nivolumab

3. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time between the date of randomization and the date of death due to any cause. Participants who do not have a date of death will be censored on the last date for which a participant was known to be alive.
Time Frame: From date of randomization to date of death (Up to 37 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 391 | 392
Months | 29.67 [22.14 to NA] — insufficient number of participants with events | 28.88 [21.32 to NA] — insufficient number of participants with events
Statistical Analysis 1: Comparison: Bempegaldesleukin + Nivolumab vs Nivolumab; Test type: Superiority — Bempegaldesleukin+Nivolumab over Nivolumab; p = 0.6361, Log Rank; 2-sided p-value. Boundary for statistical significance p-value < 0.00071; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.72 to 1.22] — Stratified Cox proportional hazard model. Hazard Ratio is NKTR-214 + Nivolumab over Nivolumab

4. Secondary Outcome: Clinical Benefit Rate (CBR) Per Blinded Independent Central Review (BICR)
Description: CBR, or equivalently the disease control rate (DCR) is defined as the percentage of participants with a best overall response of complete response (CR), partial response (PR), or stable disease (SD) as assessed by blinded independent central review (BICR) using RECIST v 1.1. CR=Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions.SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: From date of randomization to disease progression (Up to 37 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 271 | 272
Percentage of participants | 56.1 [50.0 to 62.1] | 58.5 [52.4 to 64.4]

5. Secondary Outcome: Duration of Response (DoR) Per Blinded Independent Central Review (BICR)
Description: DOR is defined for participants who have a confirmed complete response (CR) or partial results (PR) as the date from first documented CR or PR using RECIST v 1.1 to the date of the documentation of disease progression per blinded independent central review (BICR) assessment or death due to any cause, whichever is earlier. CR=Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From date of randomization to disease progression, or death, whichever is earlier (Up to 37 months)
Population: All randomized participants with partial or complete response and at least 6 months of follow-up at the time point of the final objective response rate analysis. A follow-up time is defined as the time between randomization date and clinical data cut-off date.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 75 | 98
Months | 29.67 [18.89 to NA] — insufficient number of participants with events | NA [26.74 to NA] — insufficient number of participants with events

6. Secondary Outcome: Time to Objective Response (TTR) Per Blinded Independent Central Review (BICR)
Description: Time to response (TTR) is defined for participants who had a confirmed complete response (CR) or partial response (PR) as the time from the date of randomization to date of first documented CR or PR per blinded independent central review (BICR) assessment using RECIST v 1.1. CR=Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From date of randomization to disease progression (Up to 37 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: Months
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 75 | 98
Months | 2.17 [1.0 to 15.3] | 2.20 [1.2 to 15.5]

7. Secondary Outcome: Objective Response Rate (ORR) Per Investigator
Description: ORR is defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR) using RECIST v 1.1 per investigator assessment. CR=Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From date of randomization to disease progression (Up to 37 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 271 | 272
Percentage of participants | 29.2 [23.8 to 35.0] | 36.4 [30.7 to 42.4]
Statistical Analysis 1: Comparison: Bempegaldesleukin + Nivolumab vs Nivolumab; Bempegaldesleukin+Nivolumab over Nivolumab; Test type: Superiority; p = 0.0626, Stratified Cochran-Mantel-Haenszel; two-sided; Estimate of Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.48 to 1.02] — Strata adjusted odds ratio (NKTR-214 + Nivolumab over Nivolumab) using Mantel-Haenszel method

8. Secondary Outcome: Progression-free Survival (PFS) Per Investigator
Description: PFS is defined as the time between the date of randomization and the first date of documented tumor progression using RECIST v 1.1 per investigator, or death due to any cause, whichever comes first. Progressive disease (PD)=At least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From date of randomization to disease progression, or death, whichever comes first (Up to 37 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 391 | 392
Months | 4.27 [4.04 to 6.14] | 6.21 [4.60 to 10.25]
Statistical Analysis 1: Comparison: Bempegaldesleukin + Nivolumab vs Nivolumab; Test type: Superiority; p = 0.3713, Log Rank — Log-rank stratified 2-sided. Boundary for statistical significance p-value < 0.03; Hazard Ratio (HR) = 1.09, 95% CI [0.90 to 1.33] — Stratified Cox proportional hazard model. Hazard Ratio is NKTR-214 + Nivolumab over Nivolumab

9. Secondary Outcome: Clinical Benefit Rate (CBR) Per Investigator
Description: CBR, or equivalently the disease control rate (DCR) is defined as the percentage of participants with a best overall response of complete response (CR), partial response (PR), or stable disease (SD) as assessed by investigator using RECIST v 1.1. CR=Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions. SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: From date of randomization to disease progression (Up to 37 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 271 | 272
Percentage of participants | 60.5 [54.4 to 66.4] | 61.8 [55.7 to 67.6]

10. Secondary Outcome: Duration of Response (DoR) Per Investigator
Description: DOR is defined for participants who have a confirmed complete response (CR) or partial results (PR) as the date from first documented CR or PR using RECIST v 1.1 to the date of the documentation of disease progression per investigator assessment or death due to any cause, whichever is earlier. CR=Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From date of randomization to disease progression, or death, whichever is earlier (Up to 37 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 79 | 99
Months | NA [17.31 to NA] — insufficient number of participants with events | NA [21.68 to NA] — insufficient number of participants with events

11. Secondary Outcome: Time to Objective Response (TTR) Per Investigator
Description: Time to response (TTR) is defined for participants who had a confirmed complete response (CR) or partial response (PR) as the time from the date of randomization to date of first documented CR or PR per investigator assessment using RECIST v 1.1. CR=Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From date of randomization to disease progression (Up to 37 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: Months
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 79 | 99
Months | 2.14 [1.6 to 18.3] | 2.14 [1.8 to 12.2]

12. Secondary Outcome: Objective Response Rate (ORR) Per Blinded Independent Central Review (BICR) by Baseline PD-L1 Status
Description: ORR by baseline PD-L1 tumor cells expression (PD-L1 negative: <1%) vs. (PD-L1 positive: >=1%). ORR is defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR) using RECIST v 1.1 per blinded independent central review (BICR) assessment. CR=Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From date of randomization to disease progression (Up to 37 months)
Population: All randomized participants with PD-L1 data available at baseline and at least 6 months of follow-up at the time point of the final objective response rate analysis. A follow-up time is defined as the time between randomization date and clinical data cut-off date
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 242 | 248
Percentage of participants
  Participants with baseline PD-L1 expression <1%: number analyzed (Participants) | 102 | 107
  Participants with baseline PD-L1 expression <1% | 17.6 [10.8 to 26.4] | 25.2 [17.3 to 34.6]
  Participants with baseline PD-L1 expression >=1%: number analyzed (Participants) | 140 | 141
  Participants with baseline PD-L1 expression >=1% | 36.4 [28.5 to 45.0] | 47.5 [39.1 to 56.1]
Statistical Analysis 1: Comparison: Bempegaldesleukin + Nivolumab vs Nivolumab; Bempegaldesleukin+Nivolumab vs. Nivolumab (PD-L1 Negative: <1%); Test type: Superiority; Odds Ratio (OR) = 0.63, 95% CI [0.32 to 1.24] — Logistic regression model with treatment, PD-L1 Status and treatment by PD-L1 Status interaction. Responders includes CR+PR
Statistical Analysis 2: Comparison: Bempegaldesleukin + Nivolumab vs Nivolumab; Bempegaldesleukin+Nivolumab vs. Nivolumab (PD-L1 Positive: >=1%); Test type: Superiority; p = 0.9939, Stratified Cochran-Mantel-Haenszel; Interaction P-value; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.39 to 1.02] — [estimate comment as in outcome 12, analysis 1]

13. Secondary Outcome: Progression-free Survival (PFS) Per Blinded Independent Central Review (BICR) by Baseline PD-L1 Status
Description: PFS by baseline PD-L1 tumor cells expression (PD-L1 negative: <1%) vs. (PD-L1 positive: >=1%). PFS is defined as the time between the date of randomization and the first date of documented tumor progression using RECIST v 1.1 per blinded independent central review (BICR), or death due to any cause, whichever comes first. Progressive disease (PD)=At least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From date of randomization to disease progression, or death, whichever comes first (Up to 37 months)
Population: All randomized participants with PD-L1 data available at baseline
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 349 | 357
Months
  Participants with baseline PD-L1 expression <1%: number analyzed (Participants) | 156 | 163
  Participants with baseline PD-L1 expression <1% | 3.25 [2.20 to 4.24] | 2.30 [2.17 to 4.17]
  Participants with baseline PD-L1 expression >=1%: number analyzed (Participants) | 193 | 194
  Participants with baseline PD-L1 expression >=1% | 6.24 [4.47 to 10.45] | 10.51 [6.05 to 28.88]
Statistical Analysis 1: Comparison: Bempegaldesleukin + Nivolumab vs Nivolumab; Bempegaldesleukin+Nivolumab vs. Nivo (PD-L1 negative: <1%); Test type: Superiority; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.81 to 1.43] — Unstratified Hazard Ratio
Statistical Analysis 2: Comparison: Bempegaldesleukin + Nivolumab vs Nivolumab; Bempegaldesleukin+Nivolumab vs. Nivo (PD-L1 positive: >=1%); Test type: Superiority; Hazard Ratio (HR) = 1.12, 95% CI [0.83 to 1.51] — Unstratified Hazard Ratio

14. Secondary Outcome: Overall Survival (OS) by Baseline PD-L1 Status
Description: OS by baseline PD-L1 tumor cells expression (PD-L1 negative: <1%) vs. (PD-L1 positive: >=1%). OS is defined as the time between the date of randomization and the date of death due to any cause. Participants who do not have a date of death will be censored on the last date for which a participant was known to be alive.
Time Frame: From date of randomization to date of death (Up to 37 months)
Population: All randomized participants with PD-L1 data available at baseline
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 349 | 357
Months
  Participants with baseline PD-L1 expression <1%: number analyzed (Participants) | 156 | 163
  Participants with baseline PD-L1 expression <1% | 21.16 [15.51 to 26.68] | 21.13 [16.62 to NA] — insufficient number of participants with events
  Participants with baseline PD-L1 expression >=1%: number analyzed (Participants) | 193 | 194
  Participants with baseline PD-L1 expression >=1% | NA [29.67 to NA] — insufficient number of participants with events | NA [28.88 to NA] — insufficient number of participants with events
Statistical Analysis 1: Comparison: Bempegaldesleukin + Nivolumab vs Nivolumab; Bempegaldesleukin+Nivolumab vs. Nivo (PD-L1 negative: <1%); Test type: Superiority; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.66 to 1.40] — Unstratified Hazard Ratio
Statistical Analysis 2: Comparison: Bempegaldesleukin + Nivolumab vs Nivolumab; Bempegaldesleukin+Nivolumab vs. Nivo (PD-L1 positive: >=1%); Test type: Superiority; Hazard Ratio (HR) = 0.88, 95% CI [0.58 to 1.33] — Unstratified Hazard Ratio

15. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with any grade adverse events (AEs) including treatment-related AEs, AEs leading to discontinuation of any drug, serious adverse events (SAEs), treatment-related SAEs, and deaths from first dose to 30 days post last dose. An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 30 days post last dose (Average of 11 months and a maximum up to 26 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 387 | 382
Participants
  AEs | 378 | 364
  Drug-related AEs | 351 | 281
  SAEs | 132 | 130
  Drug-related SAEs | 57 | 32
  AEs leading to discontinuation of any Drug | 65 | 56
  Deaths | 21 | 21

16. Secondary Outcome: Number of Participants With On-Treatment Laboratory Parameters That Worsened Relative to Baseline
Description: Number of participants with on-treatment laboratory parameters that worsened relative to baseline. Parameters include hematology, chemistry, liver function, and renal function using worst grade (grade 1-4 and grade 3-4) per national cancer institute (NCI) common terminology criteria for adverse events (CTCAE) v5 criteria.
  Grade 1=Mild event Grade 2=Moderate event Grade 3=Severe event Grade 4=Life threatening event
Time Frame: From first dose to 100 days post last dose (Average of 13 months and a maximum up to 28 months)
Population: All treated participants with laboratory baseline measures
Measure: Count of Participants; unit: Participants
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
Number analyzed (Participants) | 383 | 380
Participants
  Hemoglobin decreased grade 1-4: number analyzed (Participants) | 380 | 371
  Hemoglobin decreased grade 1-4 | 194 | 173
  Hemoglobin decreased grade 3-4: number analyzed (Participants) | 380 | 371
  Hemoglobin decreased grade 3-4 | 17 | 22
  Platelet count decreased grade 1-4: number analyzed (Participants) | 380 | 371
  Platelet count decreased grade 1-4 | 36 | 41
  Platelet count decreased grade 3-4: number analyzed (Participants) | 380 | 371
  Platelet count decreased grade 3-4 | 2 | 6
  Leukocytes decreased grade 1-4: number analyzed (Participants) | 380 | 371
  Leukocytes decreased grade 1-4 | 29 | 46
  Leukocytes decreased grade 3-4: number analyzed (Participants) | 380 | 371
  Leukocytes decreased grade 3-4 | 2 | 2
  Lymphocytes (absolute) decreased grade 1-4 | 304 | 194
  Lymphocytes (absolute) decreased grade 3-4 | 199 | 30
  Absolute Neutrophil count decreased grade 1-4: number analyzed (Participants) | 380 | 370
  Absolute Neutrophil count decreased grade 1-4 | 71 | 31
  Absolute Neutrophil, count decreased grade 3-4: number analyzed (Participants) | 380 | 370
  Absolute Neutrophil, count decreased grade 3-4 | 8 | 2
  Neutrophils (absolute) decreased grade 1-4: number analyzed (Participants) | 380 | 370
  Neutrophils (absolute) decreased grade 1-4 | 57 | 29
  Neutrophils (absolute) decreased grade 3-4: number analyzed (Participants) | 380 | 370
  Neutrophils (absolute) decreased grade 3-4 | 10 | 2
  Alkaline Phosphatase increased grade 1-4: number analyzed (Participants) | 378 | 367
  Alkaline Phosphatase increased grade 1-4 | 96 | 90
  Alkaline Phosphatase increased grade 3-4: number analyzed (Participants) | 378 | 367
  Alkaline Phosphatase increased grade 3-4 | 2 | 6
  Aspartate Aminotransferase increased grade 1-4: number analyzed (Participants) | 378 | 371
  Aspartate Aminotransferase increased grade 1-4 | 96 | 115
  Aspartate Aminotransferase increased grade 3-4: number analyzed (Participants) | 378 | 371
  Aspartate Aminotransferase increased grade 3-4 | 9 | 17
  Alanine Aminotransferase increased grade 1-4: number analyzed (Participants) | 379 | 371
  Alanine Aminotransferase increased grade 1-4 | 104 | 132
  Alanine Aminotransferase increased grade 3-4: number analyzed (Participants) | 379 | 371
  Alanine Aminotransferase increased grade 3-4 | 11 | 13
  Bilirubin, total increased grade 1-4: number analyzed (Participants) | 376 | 369
  Bilirubin, total increased grade 1-4 | 36 | 46
  Bilirubin, total increased grade 3-4: number analyzed (Participants) | 376 | 369
  Bilirubin, total increased grade 3-4 | 2 | 4
  Creatinine increased grade 1-4: number analyzed (Participants) | 378 | 369
  Creatinine increased grade 1-4 | 81 | 94
  Creatinine increased grade 3-4: number analyzed (Participants) | 378 | 369
  Creatinine increased grade 3-4 | 2 | 6
  Amylase increased grade 1-4: number analyzed (Participants) | 306 | 309
  Amylase increased grade 1-4 | 51 | 78
  Amylase increased grade 3-4: number analyzed (Participants) | 306 | 309
  Amylase increased grade 3-4 | 3 | 6
  Lipase, total increased grade 1-4: number analyzed (Participants) | 354 | 347
  Lipase, total increased grade 1-4 | 90 | 126
  Lipase, total increased grade 3-4: number analyzed (Participants) | 354 | 347
  Lipase, total increased grade 3-4 | 17 | 17
  Hypernatremia grade 1-4: number analyzed (Participants) | 379 | 371
  Hypernatremia grade 1-4 | 29 | 47
  Hypernatremia grade 3-4: number analyzed (Participants) | 379 | 371
  Hypernatremia grade 3-4 | 2 | 0
  Hyponatremia grade 1-4: number analyzed (Participants) | 379 | 371
  Hyponatremia grade 1-4 | 112 | 123
  Hyponatremia grade 3-4: number analyzed (Participants) | 379 | 371
  Hyponatremia grade 3-4 | 6 | 11
  Hyperkalemia grade 1-4: number analyzed (Participants) | 378 | 370
  Hyperkalemia grade 1-4 | 91 | 85
  Hyperkalemia grade 3-4: number analyzed (Participants) | 378 | 370
  Hyperkalemia grade 3-4 | 9 | 6
  Hypokalemia grade 1-4: number analyzed (Participants) | 378 | 370
  Hypokalemia grade 1-4 | 32 | 51
  Hypokalemia grade 3-4: number analyzed (Participants) | 378 | 370
  Hypokalemia grade 3-4 | 5 | 2
  Hypercalcemia grade 1-4: number analyzed (Participants) | 373 | 370
  Hypercalcemia grade 1-4 | 45 | 45
  Hypercalcemia grade 3-4: number analyzed (Participants) | 373 | 370
  Hypercalcemia grade 3-4 | 1 | 0
  Hypocalcemia grade 1-4: number analyzed (Participants) | 373 | 370
  Hypocalcemia grade 1-4 | 78 | 82
  Hypocalcemia grade 3-4: number analyzed (Participants) | 373 | 370
  Hypocalcemia grade 3-4 | 5 | 0
  Hypoglycemia grade 1-4: number analyzed (Participants) | 375 | 367
  Hypoglycemia grade 1-4 | 42 | 39
  Hypoglycemia grade 3-4: number analyzed (Participants) | 375 | 367
  Hypoglycemia grade 3-4 | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) are collected from first dose to 100 days post last dose (Average of 13 months and a maximum up to 28 months). Participants were assessed for All-cause mortality from their date of randomization to study completion date (Up to approximately 66 months).
Description: The number at Risk for All-Cause Mortality=All randomized participants. The number at Risk for SAEs and Other AEs=All treated participants.
Arm/Group | Bempegaldesleukin + Nivolumab | Nivolumab
All-Cause Mortality (participants affected / at risk) | 170/391 | 173/392
Serious Adverse Events (participants affected / at risk) | 161/388 | 172/382
Other Adverse Events (participants affected / at risk) | 357/388 | 336/382
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bempegaldesleukin + Nivolumab (N=388) | Nivolumab (N=382)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Eosinophilia (Blood and lymphatic system disorders) | 3 | 0
Lymph node haemorrhage (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocarditis (Cardiac disorders) | 3 | 4
Myopericarditis (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Thyroiditis (Endocrine disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 3
Autoimmune colitis (Gastrointestinal disorders) | 3 | 2
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 2 | 3
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 6
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 2 | 2
Immune-mediated pancreatitis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
Death (General disorders) | 1 | 1
Drowning (General disorders) | 1 | 0
Face oedema (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 4
General physical health deterioration (General disorders) | 4 | 3
Hanging (General disorders) | 1 | 0
Implant site haemorrhage (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 4
Sudden death (General disorders) | 0 | 2
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 1
Contrast media allergy (Immune system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 5
COVID-19 pneumonia (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 2 | 1
Cystitis (Infections and infestations) | 0 | 1
Cystitis klebsiella (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Klebsiella urinary tract infection (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 8
Pneumonia aspiration (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 4
Septic shock (Infections and infestations) | 1 | 1
Severe acute respiratory syndrome (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 3 | 0
Soft tissue infection (Infections and infestations) | 1 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tonsillitis bacterial (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 1 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 1 | 1
Lipase increased (Investigations) | 0 | 3
Liver function test increased (Investigations) | 1 | 1
Lymph node palpable (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Morphoea (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 37 | 40
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 7 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Encephalitis autoimmune (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 3
Myasthenia gravis (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 1 | 4
Spinal cord compression (Nervous system disorders) | 1 | 4
Syncope (Nervous system disorders) | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Adjustment disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 3
Autoimmune nephritis (Renal and urinary disorders) | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Testicular mass (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epiglottic polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Sarcoid-like reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 2
Ischaemia (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bempegaldesleukin + Nivolumab (N=388) | Nivolumab (N=382)
Anaemia (Blood and lymphatic system disorders) | 61 | 63
Eosinophilia (Blood and lymphatic system disorders) | 60 | 7
Hyperthyroidism (Endocrine disorders) | 49 | 28
Hypothyroidism (Endocrine disorders) | 74 | 52
Abdominal pain (Gastrointestinal disorders) | 33 | 34
Abdominal pain upper (Gastrointestinal disorders) | 29 | 16
Constipation (Gastrointestinal disorders) | 39 | 51
Diarrhoea (Gastrointestinal disorders) | 96 | 80
Dry mouth (Gastrointestinal disorders) | 21 | 13
Nausea (Gastrointestinal disorders) | 113 | 67
Vomiting (Gastrointestinal disorders) | 64 | 37
Asthenia (General disorders) | 68 | 42
Chills (General disorders) | 36 | 5
Face oedema (General disorders) | 20 | 0
Fatigue (General disorders) | 128 | 104
Influenza like illness (General disorders) | 71 | 9
Oedema peripheral (General disorders) | 40 | 30
Pyrexia (General disorders) | 147 | 39
COVID-19 (Infections and infestations) | 32 | 31
Upper respiratory tract infection (Infections and infestations) | 9 | 20
Infusion related reaction (Injury, poisoning and procedural complications) | 48 | 15
Alanine aminotransferase increased (Investigations) | 31 | 39
Amylase increased (Investigations) | 20 | 29
Aspartate aminotransferase increased (Investigations) | 26 | 34
Blood alkaline phosphatase increased (Investigations) | 10 | 20
Blood creatine phosphokinase increased (Investigations) | 23 | 38
Blood creatinine increased (Investigations) | 20 | 28
Lipase increased (Investigations) | 22 | 37
Weight decreased (Investigations) | 16 | 22
Decreased appetite (Metabolism and nutrition disorders) | 68 | 35
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 28
Hyponatraemia (Metabolism and nutrition disorders) | 15 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 99 | 67
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 47
Myalgia (Musculoskeletal and connective tissue disorders) | 55 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 | 36
Dizziness (Nervous system disorders) | 38 | 20
Headache (Nervous system disorders) | 64 | 56
Insomnia (Psychiatric disorders) | 31 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 53 | 45
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 31
Dry skin (Skin and subcutaneous tissue disorders) | 30 | 14
Erythema (Skin and subcutaneous tissue disorders) | 28 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 121 | 80
Rash (Skin and subcutaneous tissue disorders) | 108 | 63
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 30 | 18
Vitiligo (Skin and subcutaneous tissue disorders) | 35 | 34
Hypertension (Vascular disorders) | 27 | 34
Hypotension (Vascular disorders) | 33 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT03635983/Prot_SAP_000.pdf